CLINICAL TRIAL: NCT06932432
Title: Using Ecological Momentary Assessment to Develop an Adaptive Psychological Intervention for Young Adults With Chronic Pain
Status: Recruiting | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Caitlin Murray, Assistant Professor, Seattle Children's Hospital
Other Study IDs: K23AT012901 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain
Keywords: EMA study; childhood onset chronic pain; Young adult; Cannabis use; Real-time predictors; Health outcomes
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to determine real-time contextual vulnerabilities associated with pain in young adults to inform ideal treatment targets for a just-in-time adaptive intervention (JITAI). The main question it aims to answer is:

-What contextual factors and vulnerabilities will predict momentary, next-day, and weekly pain severity? 50 young adults, ages 18-25 with a diagnosis of childhood-onset primary chronic pain, will complete 1) baseline questionnaires on REDCap to collect data on sociodemographics, medical history and treatment, psychological health (i.e., current mood symptoms and previous psychiatric conditions/treatment), and pain (e.g., duration, location) and 2) a 28-day EMA via mobile app to collect survey data on dynamic factors.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-25
* diagnosis of childhood-onset chronic pain who were seen for an initial evaluation at Seattle Children's Hospital outpatient specialty clinics.

Exclusion Criteria:

* not fluent in English
* does not have regular access to the internet and access to a smartphone device (to complete EMA questions)
* presence of chronic disease or serious medical illness (e.g., arthritis, cancer, diabetes)
* serious cognitive impairment or developmental disorder (e.g., autism, intellectual disability)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Seattle Children's Hospital outpatient specialty clinics
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Momentary Pain intensity | Three times a day for 28 days
  One item from the Brief Pain Inventory will assess momentary pain intensity (yes/no), followed by "How much pain do you feel on average?" (11-point NRS)
Momentary Pain interference | Three times a day for 28 days
  Two items from the Brief Pain Inventory will assess pain interference with enjoyment in life, and general activity. Higher scores indicate more interference.

OTHER OUTCOMES:
Nightly sleep quality | Once a day for 28 days (morning)
  1-item from from the Insomnia Severity Index, "How would you rate the quality of your sleep last night?" will be rated on an 11-point NRS. 10 is equivalent to extremely good sleep and 0 indicates extremely poor sleep.
Momentary Social Company | Three times per day for 28 days
  2-items to collect, "Was anyone with you right before you received this survey?" and "Who were you with right before you received this survey?"
Momentary Location | Three times a day for 28 days
  One-item question to collect "Where were you right before receiving this survey?" in addition to GPA data with minute-to-minute mobility patterns collected via the Pathverse app
Momentary Fear | Three times a day for 28 days
  Two-items to assess fear associated with pain. Ratings of 0 indicate not at all and ratings of 4 indicate all the time
Momentary Positive and Negative Mood | Three times a day for 28 days
  Ten items from the Positive and Negative Affect Schedule will measure the extent to which a positive or negative feeling is experienced on a 5-point likert scale. 1 represents 'very slightly or not at all' and 5 indicates 'extremely'.
Momentary Pain Catastrophizing | Three times a day for 28 days
  Three items from the Pain Catastrophizing Scale will assess the extent of catastrophic thinking due to pain. Higher scores are associated with higher amounts of pain catastrophizing.
Momentary Pain Severity | Three times a day for 28 days
  Three items from the Brief Pain Inventory will measure pain intensity and pain interference on an 11-point numeric rating scale. 10 indicates 'pain as bad as you can imagine' and 'completely interferes'.
Daily Self-compassion | Once a day for 28 days (evening)
  Two items, to assess how kind oneself has been to others and oneself in the past 24 hours. A rating of 0 indicates, 'not at all', and a rating of 10 means 'very much so'.
Daily Mental Defeat | Once a day for 28 days (evening)
  One item to assess "Over the past 24 hours, how much has your pain brought back memories of times when you felt your pain had taken over your life?" Response options use a 0 through 10 numeric rating scale, 0 indicates 'not at all' and 10 indicates 'Very much so'.
Daily Substance Use | Once a day for 28 days (evening)
  One item to gather what substances were used within the last 24 hours. Response options include: Alcohol, Tobacco, Marijuana, Other (please specify), None of the above.
Daily Pain Coping | Once a day for 28 days (evening)
  One item to assess pain coping strategies used in the last 24 hours. Response options include: Distracted myself (e.g., hobbies, fun activities, talk with friends), Tried to relax, Looked for support from someone (talk on the phone, spend time), Didn't let my pain get me down, Still worked to accomplish my goals, Used cold or heat compresses, Drank alcohol, Used a drug, Just accepted my pain, Other (please specify), Nothing
Daily Pain Medication Use | Once a day for 28 days (evening)
  Three items to assess treatments or medications received for pain in the past 24 hours
Daily Activity Patterns | Once a day for 28 days (evening)
  Three items to measure activity patterns over the past 24 hours. Response options use a likert scale, 0 meaning 'not at all' and 4 indicating 'all the time'.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No